CLINICAL TRIAL: NCT00785005
Title: Exercise-related Perceived Rate of Exertion at Steady-State Workloads (ExPRESS) in Type 2 Diabetes Mellitus
Brief Title: What Makes Exercise Feel More Difficult to Women With and Without Type 2 Diabetes
Acronym: ExPRESS
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0849
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Exercise; Women; Research; Bike; Type; Control; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity; Limb-girdle muscular dystrophy, type 2C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the first visit, blood will be drawn for measurements of overall health (complete blood count and comprehensive metabolic panel), glucose and insulin levels, lipid levels, plasma FSH concentration, and HbA1C.
  On two separate visits, blood samples will be drawn from a warmed IV site to measure muscle metabolites which change with exercise (e.g., glucose, calcium, lactate, H+, K+, and HCO3-) and may be associated with muscle pain or fatigue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Females with Type 2 Diabetes
- 2: Females without Type 2 Diabetes

SUMMARY:
Given that sedentary behavior is associated with T2DM, the purpose of this study is to evaluate whether subjects with T2DM have a significant disincentive to performing exercise (due to greater perceived effort) . This study will prospectively compare the perceived exercise effort between T2DM and non-diabetic women while adjusting for potential confounders including baseline physical activity. This study will also assess whether perception of effort is associated with physiologic parameters related to exercise effort. Finally, we have 3 hypothesis-generating exploratory aims designed to screen for additional psychological and physiologic parameters that may increase perceived effort in those with T2DM.

Hypothesis 1: At the same absolute workload (e.g., 30 watts) and the same relative workloads, it is a greater effort for women with T2DM to exercise than for non-diabetic women.

Specific Aim 1: To determine differences in subjective perceived effort of bicycle exercise at low-to-moderate workloads in sedentary women with Type 2 Diabetes Mellitus (T2DM) vs. non-diabetic sedentary women.

Hypothesis 2: There will be a significant association between RPE and the physiologic measures related to work intensity (e.g., relative work intensity and tau2).

Specific Aim 2: In the same populations as SA1, to determine the strength of association during bicycle exercise between subjective perceived effort and physiologic measures related to work intensity.

Exploratory Aims:

Exploratory Aim 1: In the T2DM group described in SA1, to determine the strength of association during bicycle exercise between subjective effort and additional physiologic measures

Exploratory Aim 2: In the T2DM group described in SA1, to determine the strength of association during bicycle exercise between subjective effort and psychologic measures related to perception of effort.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women not participating in a regular exercise program (> one bout of exercise per week)
* If subject has diabetes, must be uncomplicated T2DM and < 25 years since T2DM diagnosis
* Ages of 50-70 years
* BMI of 25-35
* Subjects can only be taking the following oral hypoglycemic drugs: metformin, sulfonylureas or sitagliptin. Use of insulin or other oral hypoglycemic medications is not allowed.
* Persons with T2DM will be accepted for study only if they have total glycosylated hemoglobin levels (HbA1C) <8% (adequate control) on therapy.
* Control subjects must have HbA1C < 5.5% and a fasting blood glucose of <100 mg/dl suggesting no significant insulin resistance.
* All women must be post-menopausal, documented by menstrual history and follicle stimulating hormone (FSH) level.
* Current smokers will be excluded since smoking can impair CV exercise performance but people who have quit smoking for at least 1 year will be accepted for study.
* Absence of comorbid conditions will be confirmed by history, physical examination and laboratory testing.

Exclusion Criteria:

* In general, people will be excluded with any condition which could limit exercise performance.
* Persons with clinically evident distal symmetrical neuropathy, determined by evaluation of symptoms (numbness, paresthesia) and signs (elicited by vibration, pinprick, light touch, ankle jerks), will be excluded from further study as neuropathy may limit exercise performance.
* Persons with autonomic dysfunction (>20 mm fall in upright BP without a change in heart rate) will be excluded as well, due to associated limitations of exercise performance.
* Persons will be excluded if they have evidence of heart disease by history (Prior heart attack or bypass surgery, heart failure, or significant valvular disease) or abnormal resting electrocardiogram (EKG) consistent with prior infarct or latent ischemia (unless cardiovascular stress imaging or catheterization shows they do not have coronary artery disease). We will also exclude subjects with left or right bundle branch block on resting EKG (precludes recognition of ischemic EKG changes with exercise) or abnormal exercise EKG (> 1 mm ST segment depression 80 msec out in the ST segment for 3 consecutive beats).
* Persons with angina or any other exercise-limiting cardiovascular, pulmonary or musculoskeletal symptoms will be excluded as well.
* Presence of systolic blood pressure >150 at rest or >250 with exercise or diastolic pressure >95 at rest or >105 with exercise are also grounds for exclusion.
* Subjects with proteinuria (urine protein >200 mg/dl) or a creatinine > 2 mg/dl, suggestive of renal disease will be excluded.
* Subjects with total cholesterol >220 mg/dl, low density lipoprotein > 130 mg/dl, or triglycerides > 250 mg/dl will be excluded given the potential insulin resistance and endothelial dysfunction associated with these cholesterol parameters.
* Subjects taking the following medications will be excluded: insulin, oral hypoglycemic agents other than those stated in inclusion criteria, estrogen-containing hormone replacement therapy including the "estring".
* Control subjects who have an immediate family member with type 2 diabetes will be excluded.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-five sedentary post-menopausal women with uncomplicated T2DM (of duration ≤ 10 years) between the ages of 50-70 and twenty-five sedentary non-diabetic post-menopausal women between the ages of 50-70 will be recruited.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Huebschmann, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Huebschmann AG, Kohrt WM, Herlache L, Wolfe P, Daugherty S, Reusch JE, Bauer TA, Regensteiner JG. Type 2 diabetes exaggerates exercise effort and impairs exercise performance in older women. BMJ Open Diabetes Res Care. 2015 Sep 30;3(1):e000124. doi: 10.1136/bmjdrc-2015-000124. eCollection 2015. PMID 26464803